CLINICAL TRIAL: NCT01275898
Title: Assessing Cerebral Oxygenation During Different Surgical Procedures - Comparison of INVOS and ForeSight Cerebral Oximeter
Brief Title: Comparison of INVOS and FORE SIGHT Cerebral Oximeter
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Other Study IDs: CLS_001
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2011-08-05 (Estimated); Status verified 2010-03

CONDITIONS: Changes in Cerebral Oxygenation During Different Patient Positioning; Coparison of Two Cerebral Oximeters
Keywords: NIRS; cerebral oxygenation

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Beach chair: Patients scheduled for surgical procedure in beach chair position (Shoulder surgery)
- Sitting position: Patients scheduled for surgical procedure in sitting position (Neurosurgery)
- Head down position: Patients scheduled for surgical procedure in head down position (daVinci robotic surgery)
- Prone position: Patients scheduled for surgical procedure in prone position

SUMMARY:
Cerebral oxygenation can be monitored using near infrared spectroscopy. Different devices are available to assess cerebral oxygenation noninvasively. Beach chair position is assumed to influence cerebral oxygenation. Litte is known about the influence of prone position and head down position on cerebral oxygenation. The investigators hypothesize that these positions influence cerebral oxygenation. Further the investigators presume that the two cerebral oximeters INVOS and ForeSight provide comparable oxygenation data.

ELIGIBILITY:
Inclusion Criteria:

age >18 and <80 years written informed consent

Exclusion Criteria:

cerebrovascular disease coronary heart disease severe organ failure hemoglobin < 10mg/dl injury of forehead pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for surgical intervention in beach chair position, prone position and head down position
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2010-04

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Anaesthesiologie Universitätsmedizin Mainz, Mainz, Germany

REFERENCES:
- [Derived] Schramm P, Tzanova I, Hagen F, Berres M, Closhen D, Pestel G, Engelhard K. Cerebral oxygen saturation and cardiac output during anaesthesia in sitting position for neurosurgical procedures: a prospective observational study. Br J Anaesth. 2016 Oct;117(4):482-488. doi: 10.1093/bja/aew250. Epub 2016 Oct 17. PMID 28077536
- [Derived] Closhen D, Engelhard K, Dette F, Werner C, Schramm P. Changes in cerebral oxygen saturation following prone positioning for orthopaedic surgery under general anaesthesia: a prospective observational study. Eur J Anaesthesiol. 2015 Jun;32(6):381-6. doi: 10.1097/EJA.0000000000000259. PMID 25828385
- [Derived] Closhen D, Treiber AH, Berres M, Sebastiani A, Werner C, Engelhard K, Schramm P. Robotic assisted prostatic surgery in the Trendelenburg position does not impair cerebral oxygenation measured using two different monitors: A clinical observational study. Eur J Anaesthesiol. 2014 Feb;31(2):104-9. doi: 10.1097/EJA.0000000000000000. PMID 24225725